CLINICAL TRIAL: NCT05276635
Title: Effectiveness of Emotional Freedom Techniques vs Sleep Hygiene Education Group Therapy (SHE) in Management of Sleep Disorders Among Elderly
Brief Title: Sleep Disorder Manage in Emotional Freedom Techniques vs Sleep Hygiene Education Group Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matrouh University (Other)
Collaborators: Beni-Suef University (Other); University of Bisha (Other); Suez Canal University (Other)
Responsible Party: Principal Investigator, Nancy Elsakhy, Lecturer of Gerontological Nursing, Matrouh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0305317/2021
Record Dates: First submitted 2022-02-19; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Sleep Disorder; Sleep Disorder in Elderly; Sleep Disorder, Mental Health; Sleep Disorders, Physical Health; Sleep Disorder; Insomnia Type; Sleep Hygiene
Keywords: Emotional Freedom Techniques; Sleep Hygiene Education Geriatric; Sleep Disorders; Elderly
MeSH Terms: conditions — Sleep Wake Disorders; Psychological Well-Being; Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: An open-label randomized controlled trial design was utilized in this study. It was open-label because the type of intervention could not be concealed to participants or researchers.
Who Masked: Outcomes Assessor
Masking Description: This open-label randomised controlled trial study was conducted at Elabbasia Mental Hospital and Osana family wellness elderly nursing home at Maadi, Cairo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (EFT) (Other): had a form of Emotional Freedom Techniques (EFT) adapted for use with insomnia (EFT-I)
  Interventions: Behavioral: Emotional Freedom Techniques (EFT)
- Sleep Hygiene Education (SHE) intervention group (Active Comparator): received a Sleep Hygiene Education (SHE) intervention
  Interventions: Behavioral: The Sleep Hygiene Education (SHE)

INTERVENTIONS:
Behavioral: The Sleep Hygiene Education (SHE) — Patients were randomized into two equal groups of 30 participants each. One group received a Sleep Hygiene Education (SHE) intervention
  Other Names: Emotional Freedom Techniques (EFT)
  Arms: Sleep Hygiene Education (SHE) intervention group
Behavioral: Emotional Freedom Techniques (EFT) — 30 participants had a form of Emotional Freedom Techniques (EFT) adapted for use with insomnia (EFT-I).
  Arms: Control (EFT)

SUMMARY:
Sleep disorders are common among elderly persons, with deleterious effects on their physical and mental health. Many approaches are used to manage such disorders. Aim of the study: To compare the Emotional Freedom Techniques-Insomnia (EFT-I) and Sleep Hygiene Education (SHE) group therapy as two treatments for insomnia in a geriatric population when delivered, and their effects on sleep quality, depression, and life satisfaction.

DETAILED DESCRIPTION:
Background: Sleep disorders are common among elderly persons, with deleterious effects on their physical and mental health. Many approaches are used to manage such disorders. Aim of the study: To compare the Emotional Freedom Techniques-Insomnia (EFT-I) and Sleep Hygiene Education (SHE) group therapy as two treatments for insomnia in a geriatric population when delivered, and their effects on sleep quality, depression, and life satisfaction. Participants and methods: This open-label randomized controlled trial study was conducted at Elabbasia Mental Hospital and Osana family wellness elderly nursing home at Maadi, Cairo. It included 60 elderly patients suffering insomnia sleep problem randomized into two equal groups: one group received a Sleep Hygiene Education (SHE) intervention, the other had a form of Emotional Freedom Techniques (EFT) adapted for use with insomnia (EFT-I). A self-administered questionnaire with tools for sleep quality (Pittsburgh Sleep Quality Index [PSQI]), depression, and life satisfaction was used to collect data. The fieldwork was from January to March 2021.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering insomnia sleep problem
* Age equal or more than 60 years

Exclusion Criteria:

* Those having major physical or psychiatric ailments or being on medication affecting their sleep were excluded
* These involved those history of epilepsy, seizures, or dementia, current alcohol or substance abuse/dependence (must have >90 days of sobriety), night shift workers, as well as those unable to complete the study questionnaires and psychological tests.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male gender, represented by 17(56.7%) and 16 (53.3%) in the EFT and Sleep hygiene groups; respectively. However, Female participants was 13 (43.3%) and 14(46.7%) in both groups respectively.
Enrollment: 60 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
poor quality sleep (PSQI) | The tool filling can be completed in 5-10 minutes
  The tool consists of 19 items from which seven components covering different aspects of sleep are computed to produce one composite global score. These are sleep latency asking about how long it takes to fall asleep, sleep duration, habitual sleep efficiency measuring the percentage of sleep time of total bedtime, sleep disturbances, use of sleeping medication, daytime dysfunction, in addition to overall subjective sleep quality. Each item is weighted on a 0-3 interval scale, with a higher score indicating worse quality. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. For categorical analysis, the total score in dichotomized into good sleep quality (total score <=5), and poor sleep quality (total score >5) [15].
Geriatric Depression Scale (GDS-15) | The tool filling can be completed in 5-10 minutes
  The Geriatric Depression Scale 15-item version. It also helps in the assessment of the severity of these symptoms and in treatment follow-up. we applied the modifed 15-question shorter version as proposed by Sheikh and Yesavage 1986, and its validity was put in evidence. The tool has 15 items such as: "Are you basically satisfied with your life?", "Do you often get bored?"," Do you feel happy most of the time?", "Do you think that most people are better off than you are?". The response to each item is either Yes or No. These are scored 1 and zero respectively. The scoring was reversed for positive items so that a higher score indicates more severe depression. The scores of the items are summed-up giving a total score ranging from 0 to 15. For categorical analysis, the total score in dichotomized into: no depression (total score <=5), and depression (total score >5). The validated Arabic version of this tool was used in the present study.
Satisfaction with Life (SWL) scale | The tool filling can be completed in 5-10 minutes
  The third tool was the Satisfaction with Life (SWL) scale. This tool was developed by Diener et al. [23], to assess a person's to overall subjective feeling of satisfaction with his/her life. The tool consists of five items such as "In most ways my life is close to my ideal", "If I could live my life over, I would change almost nothing." The responses are on a 7-point Likert type scale ranging from "strongly disagree' to "strongly agree." These are scored from one to seven. The scores of the items are summed-up giving a total score ranging from 5 to 35. For categorical analysis, the total score in dichotomized into: dissatisfied (total score 5-20), and satisfied (total score 21-35). Research demonstrated high tool validity and reliability [24, 25]. Arabic version of this tool was used in the present study.
  The validity of this Scale according to Cronbach's alpha was 0.87
Pilot study | two months
  A pilot study was conducted on six patients representing 10% of computed sample size to test the clarity of the data collection form and the feasibility of the research process. Needed modifications were carried out based on the results of the pilot study, and the tool was finalized accordingly. The patients involved in the pilot were excluded from the study to avoid contamination of the study sample.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Matrouh University, Marsá Maţrūḩ, Egypt

IPD SHARING:
Plan to Share IPD: No